CLINICAL TRIAL: NCT06383065
Title: Early Effects of Physiotherapy Program Applied Before and After Bariatric Surgery on Respiratory Function, Respiratory Muscle Strength and Functional Capacity in Patients With Type 2 Diabetes
Brief Title: Respiratory Physiotherapy in Type 2 Diabetes and Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Melis Bagkur, assist prof, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YDU/2020/76-1007
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; Bariatric Surgery Candidate
Keywords: Diabetes Mellitus; Respiratory Muscles; Bariatric Surgery; Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): In the IMT group, only IMT will be applied on the first day before surgery, and the hospital routine exercise program will be applied in addition to IMT treatment from the first day to the fourth postoperative day.
  Interventions: Other: IMT Group
- Control Group (No Intervention): Individuals in the control group will be applied only the hospital routine exercise program in the postoperative period.

INTERVENTIONS:
Other: IMT Group — Inspiratory muscle training involves breathing exercises using a pressure threshold device to strengthen the muscles involved in breathing in.
  Arms: IMT group

SUMMARY:
The aim of this study is to investigate the early effects of Inspiratory Muscle Training (IMT) applied before and after bariatric surgery on respiratory function, respiratory muscle strength and functional capacity in individuals with type 2 diabetes.

The study will be conducted with 40 individuals with type 2 diabetes aged between 25-65. Individuals will be randomly assigned to the IMT (trained at 30% of maximum inspiratory pressure with an IMT threshold device) and control group. As measurement parameters, a 6-minute walk test for functional capacity, a spirometry test for respiratory function, and a portable device (Cosmed Pony FX Desktop Spirometer, USA) will be used for respiratory muscle strength. Hand grip strength will be measured with a Baseline dynamometer. All measurements will be repeated on the first day before surgery and on the fourth day before discharge after surgery.

DETAILED DESCRIPTION:
All patients will be evaluated with the same examinations on the first day before surgery and on the fourth day after surgery before discharge. Individuals in the control group will only apply the hospital routine exercise program in the postoperative period. While individuals in the IMT group will receive only IMT on the first day before surgery, they will also receive the hospital routine exercise program in addition to IMT treatment from the first day to the fourth day after surgery. During the training, the patient will undergo two 20-minute training sessions with a linear pressure resistance device, wearing a nose clip (Threshold® IMT-Health Scan Products, USA) in a sitting position (ATS/ETS, 2002). IMT training load will be adjusted according to the 30-40% pressure determined in the MIP measurement. In the postoperative period, all patients will receive incentive spirometry, breathing exercises and ambulation exercises as part of the hospital routine exercise program.

ELIGIBILITY:
Inclusion Criteria:

• Individuals with type 2 diabetes between the ages of 25 and 65 who applied to the General Surgery Department of Büyük Anadolu Hospital and underwent bariatric surgery

Exclusion Criteria:

* Individuals with a history of emergency surgery,
* Smoking,
* Exercising regularly in the last 6 months,
* Comorbidities with respiratory dysfunction,
* Pulmonary dysfunction,
* Acute COPD exacerbation were excluded from the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 5 days
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) were evaluated with a portable device (Cosmed Pony FX Desktop Spirometer, USA). MIP measurement was performed at the residual volume.
Respiratory Function | 5 days
  The respiratory function measured using a spirometer device (Cosmed Srl, Cosmed Pony Fx, Rome, Italy) consisted of physiological measurement of the volume and flow per second of the air entering and exiting the lungs of the individual during inspiration and expiration
Functional Capacity: The 6-minute walk test | 5 days
  The 6-minute walk test is a practical test that can easily be applied at the level of submaximal effort used in the evaluation of functional capacity. The test is performed indoors, in a 30-meter flat, non-slippery place with marked two ends, and where there is no material to hinder the person being tested.
Hand Grip Strength | 5 days
  Grip strength in the dominant and nondominant hand was evaluated in 'kg' using the grip hand dynamometer (Baseline Smedley, Model 12-0286, White Plains, NY, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No